CLINICAL TRIAL: NCT06979908
Title: A Clinical Study on the Efficacy and Safety of Fruquintinib in Combination With PD-1 Monoclonal Antibody and Chidamide in Refractory MSS Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Wang Chang, Director, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-Q103
Record Dates: First submitted 2025-05-09; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Fruquintinib: 5 mg, once daily, orally, on days 1-14, every 3 weeks (Q3W); Sintilimab (PD-1 inhibitor): 200 mg, once per cycle, intravenous infusion (first infusion over 60 minutes, subsequent infusions over 30-60 minutes), on day 1, Q3W; Chidamide: 30 mg, twice weekly (BIW), orally (with at least 3 days between doses, taken 30 minutes after meals).
  Interventions: Drug: Fruquintinib+Sintilimab+Chidamide

INTERVENTIONS:
Drug: Fruquintinib+Sintilimab+Chidamide — Fruquintinib: 5 mg orally once daily on days 1-14 of each 21-day cycle (Q3W).
  Sintilimab (anti-PD-1): 200 mg intravenously on day 1 of each cycle (first infusion over 60 minutes, subsequent infusions over 30-60 minutes, Q3W).
  Chidamide: 30 mg orally twice weekly (BIW; e.g., Monday & Thursday or Tuesday & Friday, with ≥3 days between doses), taken 30 minutes after meals.

SUMMARY:
This study is a single-arm, open-label, single-center clinical trial designed to evaluate the efficacy and safety of fruquintinib in combination with a PD-1 inhibitor and chidamide in patients with refractory MSS-type metastatic colorectal cancer (mCRC). A total of 46 patients are planned to be enrolled, with the primary endpoint being median progression-free survival (mPFS). Secondary endpoints include median overall survival (mOS), objective response rate (ORR), and safety.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and ability to comply with the study protocol.
* Age ≥18 years and ≤75 years.
* Histologically confirmed colorectal adenocarcinoma.
* Unresectable locally advanced, unresectable recurrent, and/or metastatic disease (i.e., advanced disease not amenable to curative treatments such as radical radiotherapy, chemoradiotherapy, and/or surgery) after failure of ≥2 prior lines of standard therapy.
* At least one measurable lesion as per RECIST v1.1.
* ECOG performance status of 0 or 1.
* Life expectancy ≥3 months.
* Adequate bone marrow, liver, and renal function:

ANC ≥1.5 × 10⁹/L (1500/µL) Platelet count ≥100 × 10⁹/L (100,000/μL) Hemoglobin ≥90 g/L (9 g/dL) For patients without liver metastases: AST/ALT ≤2.5 × ULN For patients with liver metastases: AST/ALT ≤5 × ULN Total bilirubin ≤1.5 × ULN Serum creatinine ≤1.5 × ULN and creatinine clearance ≥60 mL/min

* For women of childbearing potential (WOCBP): Negative urine or serum pregnancy test within 3 days prior to the first dose of study treatment.
* Contraception requirement: All subjects (male or female) at risk of conception must use highly effective contraception (failure rate <1% per year) throughout the treatment period and for 120 days after the last dose of study drug (or 180 days after the last dose of chemotherapy, if applicable).

Exclusion Criteria:

* Palliative radiotherapy for colorectal cancer within 4 weeks prior to initiation of study treatment.
* Use of traditional Chinese medicine (TCM) or Chinese herbal preparations for cancer control within 7 days before starting study treatment.
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.
* Other severe uncontrolled comorbidities (e.g., interstitial lung disease, epilepsy, hepatic failure, etc.).
* Current or history of autoimmune diseases or immunodeficiency disorders.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonia on screening chest CT.
* Severe chronic or active infection requiring treatment within 4 weeks prior to study treatment initiation.
* Major surgery (excluding diagnostic procedures) within 4 weeks before study treatment or anticipated need for major surgery during the study period.
* Clinically significant cardiovascular disease, including:Symptomatic congestive heart failure (CHF),Poorly controlled hypertension,Unstable angina,Arrhythmias,Myocardial infarction within 6 months,Arterial thromboembolism or pulmonary embolism within 3 months before the first dose.
* History of other malignancies (except the cancer under investigation) within 2 years prior to screening.
* Prior immune checkpoint inhibitor therapy (e.g., anti-CTLA-4, anti-PD-1, anti-PD-L1).mmunostimulatory agents (e.g., IFN, IL-2) within 4 weeks before study treatment, or 5 drug elimination half-lives (whichever is longer).
* Chemotherapy, immunotherapy (e.g., IL, IFN, thymosin), or any investigational therapy within 14 days before study treatment, or5 drug elimination half-lives (whichever is longer).
* Active or chronic infections, including:HIV-positive,Active hepatitis B (HBV) or hepatitis C (HCV), or related medical history.
* For HBV carriers (HBsAg+ or HBcAb+):HBV DNA must be ≤2.5×10³ copies/mL (or ≤500 IU/mL) or below detection limit to enroll.Antiviral therapy for HBV is mandatory throughout the study.For HCV-seropositive patients:HCV RNA must be negative or below detection limit for enrollment.
* Any other condition deemed by the investigator to increase the risk of premature study termination.
* Patients who required systemic corticosteroid therapy (>10 mg/day prednisone or equivalent) or other immunosuppressants within 14 days prior to the first dose. In the absence of active autoimmune disease, inhaled or topical corticosteroids are permitted, as well as adrenal replacement therapy at doses ≤10 mg/day prednisone equivalent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-07-22 (Estimated); Study Completion 2027-01-22 (Estimated)

PRIMARY OUTCOMES:
PFS | 24 months
  Progression-Free Survival

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China